CLINICAL TRIAL: NCT02943707
Title: Autologous Bone Marrow Stem Cells Infusion for the Treatment of Liver Diseases.
Acronym: ABMSCIFTLD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, yongping chen, Director,Clinical Research, Wenzhou Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12330000470005914R
Record Dates: First submitted 2016-10-17; First posted 2016-10-25 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Liver Diseases
Keywords: liver diseases; Bone Marrow Cell Transplantation
MeSH Terms: conditions — Liver Diseases | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment group: ABMSCi & drugs (Experimental): ABMSCi: Autologous bone marrow stem cells infusion drugs such as Ursodeoxycholic Acid tablets(UDCA), each time 150 mg, three times a day orally
  Interventions: Procedure: Autologous bone marrow stem cells infusion; Drug: drugs such as Ursodeoxycholic Acid tablets
- control group: drugs (Active Comparator): drugs such as Ursodeoxycholic Acid tablets(UDCA), each time 150 mg, three times a day orally
  Interventions: Drug: drugs such as Ursodeoxycholic Acid tablets

INTERVENTIONS:
Procedure: Autologous bone marrow stem cells infusion — Autologous bone marrow stem cells are infused into proper hepatic artery
  Other Names: ABMSCi
  Arms: treatment group: ABMSCi & drugs
Drug: drugs such as Ursodeoxycholic Acid tablets — Ursodeoxycholic Acid tablets(UDCA), each time 150 mg, three times a day orally
  Other Names: UDCA

SUMMARY:
This study evaluates the effect of autologous bone marrow stem cells infusion (ABMSCi) therapy for liver diseases.Treatment group will receive ABMSCi and drugs therapy ,while control group will only receive drugs therapy.

DETAILED DESCRIPTION:
1. Autologous bone marrow stem cells (ABMSC) mobilization and harvest For harvesting more ABMSC, ABMSC mobilization is induced by recombinant human granulocyte colony stimulating factor (rhGCSF,Gran○R), administered subcutaneously at a dose of 300μg daily for three consecutive days before bone marrow puncture.

   Bone marrow (160-200ml) of the patients is harvested from both posterior superior iliacs according to standard procedures under local anaesthesia and is collected in a plastic bag containing heparin.
2. Both treatment group and control group receive drugs therapy.
3. ABMSC separation and infusion ABMSC is separated and purified in a class 10,000 clean laboratory. After fat and bony particles are removed by filtration, collected cells are moved to a cell-processing device. The reagents adopt the method of negative cells collection. Take the cells which intended to remove as target cells, and carry out the removal step-by-step. On the basis of this method, red blood cells, blood platelets, blood plasma will be completely removed with part of white cells and lymphocytes being remarkably removed as well while all the stem cells / progenitor cells are being well retained.

   The nucleated cell (white blood cell) count of final ABMSC is measured by an automated complete blood count instrument and flow cytometry analysis. The number of mononuclear cells is counted manually under a microscope by Wright-Giemsa stain method. Cell differentiation factor 34(CD34) positive cells were determined by flow cytometry analysis.

   The time of ABMSC separation and purification is 2.5-3 hours. ABMSC is added to 10 ml saline and well mixed by shaking the vial gently. The catheter is pushed to reach the proper hepatic artery. The diameter of the catheter is 1.4mm, it is thin enough to easily been inserted to right gastric artery . The mixture of saline and ABMSC is infused into proper hepatic artery at uniform speed for about two minutes. The catheter is removed after the ABMSCi.
4. Statistical analysis - Categorical data are presented as absolute values and percentages, whereas continuous data are summarized as mean and Standard Deviation. Statistical analysis was performed using t-test for paired or unpaired samples. Time courses of measurements of liver function parameters were analyzed by repeated-measures ANOVA. The analysis is performed using the Statistic Package for Social Science (SPSS). All statistical analysis is based on two-tailed hypothesis tests with a significance level of p< 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Definite liver diseases (such as viral hepatitis, autoimmune liver diseases, fatty liver diseases, ect);
2. Active bone marrow hyperplasia showed by bone marrow biopsy before ABMSCi;
3. Age between 18 and 60 years;
4. Abnormal liver function.

Exclusion Criteria:

1. Enlisted for liver transplantation
2. Diagnosis of hepatocellular carcinoma or other cancers
3. Other severe medical disease, and acute infection
4. pregnant or nursing females,co-infections with HIV ,serious bacterial infection
5. other vital organ or system dysfunction
6. with severe complications of liver cirrhosis
7. hematological disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline alanine aminotransferase at 6 months | baseline and 6 months after treatment
  alanine aminotransferase (ALT)
Change from baseline aspartate aminotransferase at 6 months | baseline and 6 months after treatment
  aspartate aminotransferase (AST)
Change from baseline total bilirubin at 6 months | baseline and 6 months after treatment
  total bilirubin (TBil)
Change from baseline direct bilirubin at 6 months | baseline and 6 months after treatment
  direct bilirubin (DBil)
Change from baseline total bile acid at 6 months | baseline and 6 months after treatment
  total bile acid (TBA)
Change from baseline albumin at 6 months | baseline and 6 months after treatment
  albumin (ALB)
Change from baseline prothrombin time at 6 months | baseline and 6 months after treatment
  prothrombin time (PT),
Change from baseline international normalized ratio at 6 months | baseline and 6 months after treatment
  international normalized ratio (INR)
Change from baseline white blood cell at 6 months | baseline and 6 months after treatment
  white blood cell (WBC)
Change from baseline platelet at 6 months | baseline and 6 months after treatment
  platelet (PLT)

SECONDARY OUTCOMES:
Change from baseline liver density at 6 months | baseline and 6 months after treatment
  Low density, medium density, high density tested by abdominal B ultrasound/CT/MRI
Change from baseline liver size at 6 months | baseline and 6 months after treatment
  Enlarged size, normal size, shrunken size tested by abdominal B ultrasound/CT/MRI
Change from baseline spleen thickness at 6 months | baseline and 6 months after treatment
  tested by abdominal B ultrasound/CT/MRI
Incidence of adverse events that are related to treatment | baseline and 6 months after treatment
  Postoperative pyrexia, infection, liver cirrhosis, ascites, upper gastrointestinal hemorrhage, malignant tumors of liver and other organs
Number of participants that survive without developing disease | 12 months after treatment
Number of participants that survive with developing disease | 12 months after treatment
Number of participants that die after treatment | 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: yongping chen, Study Chair — First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- the First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ma XR, Tang YL, Xuan M, Chang Z, Wang XY, Liang XH. Transplantation of autologous mesenchymal stem cells for end-stage liver cirrhosis: a meta-analysis based on seven controlled trials. Gastroenterol Res Pract. 2015;2015:908275. doi: 10.1155/2015/908275. Epub 2015 Mar 15. PMID 25861263
- [Result] Xu L, Gong Y, Wang B, Shi K, Hou Y, Wang L, Lin Z, Han Y, Lu L, Chen D, Lin X, Zeng Q, Feng W, Chen Y. Randomized trial of autologous bone marrow mesenchymal stem cells transplantation for hepatitis B virus cirrhosis: regulation of Treg/Th17 cells. J Gastroenterol Hepatol. 2014 Aug;29(8):1620-8. doi: 10.1111/jgh.12653. PMID 24942592
- [Result] Peng L, Xie DY, Lin BL, Liu J, Zhu HP, Xie C, Zheng YB, Gao ZL. Autologous bone marrow mesenchymal stem cell transplantation in liver failure patients caused by hepatitis B: short-term and long-term outcomes. Hepatology. 2011 Sep 2;54(3):820-8. doi: 10.1002/hep.24434. Epub 2011 Jul 14. PMID 21608000
- [Result] Deng Q, Cai T, Zhang S, Hu A, Zhang X, Wang Y, Huang J. Autologous Peripheral Blood Stem Cell Transplantation Improves Portal Hemodynamics in Patients with Hepatitis B Virus-related Decompensated Cirrhosis. Hepat Mon. 2015 Dec 20;15(12):e32498. doi: 10.5812/hepatmon.32498. eCollection 2015 Dec. PMID 26977164
- [Result] Mohamadnejad M, Vosough M, Moossavi S, Nikfam S, Mardpour S, Akhlaghpoor S, Ashrafi M, Azimian V, Jarughi N, Hosseini SE, Moeininia F, Bagheri M, Sharafkhah M, Aghdami N, Malekzadeh R, Baharvand H. Intraportal Infusion of Bone Marrow Mononuclear or CD133+ Cells in Patients With Decompensated Cirrhosis: A Double-Blind Randomized Controlled Trial. Stem Cells Transl Med. 2016 Jan;5(1):87-94. doi: 10.5966/sctm.2015-0004. Epub 2015 Dec 10. PMID 26659833
- [Result] Chen Y, Chen S, Liu LY, Zou ZL, Cai YJ, Wang JG, Chen B, Xu LM, Lin Z, Wang XD, Chen YP. Mesenchymal stem cells ameliorate experimental autoimmune hepatitis by activation of the programmed death 1 pathway. Immunol Lett. 2014 Dec;162(2 Pt B):222-8. doi: 10.1016/j.imlet.2014.10.021. Epub 2014 Oct 28. PMID 25445618